CLINICAL TRIAL: NCT03843931
Title: A Randomized, Open Label, Parallel Group Study in Patients With Knee Osteoarthritis to Compare Intra-articular Saline Injections With Education Plus Exercise Therapy
Brief Title: Saline Injections vs Education and Exercise in Knee Osteoarthritis
Acronym: DISCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APPI2-PT-2019-01
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Exercise; Placebo; Injection
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Educational Status; Exercise; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLA:D (Active Comparator): 8 weeks of education (1 session/week for 2 weeks) and exercise therapy (2 sessions/week for 6 week)
  Interventions: Behavioral: GLA:D
- Intra-articular saline injection (Placebo Comparator): Intra-articular saline injection (5 ml of 0.9% sodium chloride) every 2 weeks over an 8-week period
  Interventions: Drug: Intra-articular saline injection

INTERVENTIONS:
Behavioral: GLA:D — The GLA:D exercise and education program is an 8-week treatment program delivered by GLA:D certified physiotherapists. It consists of 2 educational sessions over 2 weeks (1/week in week 1 and 2) and 12 exercise sessions over 6 weeks (2/week in weeks 2 thru 8) The 2 educational sessions provide knowledge of OA, treatment and self-management, with a special focus on exercise and its benefits. The exercise part lasts for 6 weeks with 2 exercise sessions per week of approximately 1 hour (12 sessions total). The exercise sessions are group based at a facility supervised by a GLA:D certified physiotherapist. The goal is the obtain muscle control and stability in situations resembling daily life and/or more strenuous activities.
  Other Names: Education and Exercise
  Arms: GLA:D
Drug: Intra-articular saline injection — Four [4] dosages of 5 ml intra-articular isotonic saline (0.9% (9 mg/mL) Sodium Chloride Injection (sterile, isotonic solution of sodium chloride and sterile water for injection)) every other week from baseline (week 1, 3, 5 and 7 = 4 injections).
  The injections will be carried out with a 21 gauge (38 mm) needle and a Luer-lock syringe under ultrasound guidance to ensure that the needle is inserted into the study knee joint cavity and document correct deposition of the bolus in the joint cavity.
  If the investigator detects presence of excessive joint fluid during the ultrasound guided preparation of the injection, this will be aspirated before injection of the saline - if possible.
  Other Names: Physiological salinated water
  Arms: Intra-articular saline injection

SUMMARY:
Knee osteoarthritis (OA) is a highly prevalent musculoskeletal condition mainly affecting older people, causing pain, physical disability, and reduced quality of life. Exercise and patient education are non-pharmacological interventions for knee OA unanimously recommended by leading international organisations and authorities based on extensive research that documents that exercise and education are superior to no-attention control groups.

In Denmark, an initiative to implement these recommendations was initiated in 2013. The initiative is called Good Life with osteoArthritis in Denmark (GLA:D) and aims at facilitating high quality care of patients with OA in the Danish population. The core components of the GLA:D program are 8 weeks of education (2 sessions) and supervised neuromuscular exercise delivered by GLA:D certified physiotherapists. The GLA:D concept has been exported to Canada, China and Australia.

While several randomised controlled trials have investigated exercise and education for knee OA none have used a placebo comparison group. The effect size of exercise plus education therapy is in line with the current theories that the contact with a caring clinician that believes in efficacy of the treatments he/she provides can result in beneficial health effects. In exercise and education programs (such as the GLA:D program) frequent and lengthy contacts with a physiotherapist are typically necessary. Hence, a significant proportion of the beneficial effects can be expected to be attributable to placebo or placebo.like effects.

In trials of intra-articular treatment of knee OA (e.g. in trials of corticosteroids, viscosupplementation, or platelet-rich-plasma) saline injections are a commonly used as placebo comparator. While saline is recognised as a pharmacologically inert agent, a recent systematic review and meta-analysis concluded that although intra-articular saline injection is often used as a "placebo" treatment in clinical trials for knee OA it can provide substantial pain relief. The effect size of saline injections is in line with the current theories that the "invasiveness" of a procedure is an important determinant for the magnitude of placebo effects.

This trial aims to compare a widely used 8-week education plus exercise program (the GLA:D program) with 4 intra-articular saline injections as treatments of knee OA symptoms. Outcomes are taken at baseline, after 8-weeks of treatment (week 9) and after additionally 4 weeks of follow-up (week 12).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years.
2. Body Mass index ≤ 35
3. A clinical diagnosis of tibiofemoral OA in the target knee according to the American College of Rheumatology (12).
4. Average knee pain in the last week during weight bearing activities of at least 4 on a 0 to 10 points scale (0=no pain; 10=worst possible pain).
5. Verification of clinical diagnosis by definite tibiofemoral OA on posterior-anterior weight bearing semi-flexed knee radiographs with severity equivalent to Kellgren and Lawrence grade 2 or more.

Exclusion Criteria:

1. Intra-articular treatments of any kind of either knee 3 months before inclusion
2. Scheduled surgery during study participation
3. Knee joint fluid aspiration within 3 month of baseline visit
4. Participation in exercise therapy within 3 months of baseline visit
5. Evidence of other inflammatory joint disease (e.g. rheumatoid arthritis or gout)
6. History of knee surgery within 12 months
7. History of arthroplasty in the target knee
8. Use of oral glucocorticoids
9. Use of synthetic or non-synthetic opioids
10. Other musculoskeletal, neurological, medical conditions precluding participation in exercise
11. Contraindications to intra-articular injections, such as wounds or skin rash over injection site.
12. Contraindications to exercise
13. Planning to start other treatment for knee OA in the study participation period
14. Regional pain syndromes
15. Generalised pain syndromes such as fibromyalgia
16. Lumbar or cervical nerve root compression syndromes
17. Any other condition or impairment that, in the opinion of the investigator, makes a potential participant unsuitable for participation or which obstruct participation, such as large knee joint effusion, uncontrolled diabetes, psychiatric disorders, or opiate dependency.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in knee pain | week 9
  Assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) pain subscale (patient-reported questionnaire).
  The KOOS pain subscale consists of 9 questions with a five-point Likert scale scoring system (ranging from 0 (least severe) to 4 (most severe)). The answers are summed and a 0-100 normalized score is calculated with 0 indicating extreme pain and 100 indicating no pain.

SECONDARY OUTCOMES:
Change from baseline in physical function | week 9 and week 12
  Assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) physical function subscale (patient-reported questionnaire)The KOOS physical function subscale consists of 17 questions with a five-point Likert scale scoring system (ranging from 0 (least severe) to 4 (most severe)). The answers are summed and a 0-100 normalized score is calculated with 0 indicating extreme functional impairment and 100 indicating no functional impairment.
Change from baseline in symptoms | week 9 and week 12
  Assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) symptoms subscale (patient-reported questionnaire) The KOOS symptoms subscale consists of 7 questions with a five-point Likert scale scoring system (ranging from 0 (least severe) to 4 (most severe)). The answers are summed and a 0-100 normalized score is calculated with 0 indicating extreme symptoms and 100 indicating no symptoms.
Change from baseline in knee related quality of life | week 9 and week 12
  Assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) knee related quality of life subscale (patient-reported questionnaire) The KOOS knee related quality of life subscale consists of 4 questions with a five-point Likert scale scoring system (ranging from 0 (least severe) to 4 (most severe)). The answers are summed and a 0-100 normalized score is calculated with 0 indicating extremely poor knee related quality of life pain and 100 indicating very good knee related quality of life .
Change from baseline in patient's global assessment of impact of osteoarthritis | week 9 and week 12
  Assessed by a 0-100 mm visual analog scale (VAS)(patient-reported questionnaire)
Number of treatment responders according to OMERACT-OARSI response criteria | week 9 and week 12
  following two conditions is observed at the post-baseline assessment:
  * In either pain (KOOS pain subscale) or function (KOOS function subscale), a high improvement in the subscale, where high improvement in a subscale is achieved if there is both a > 50% improvement from Baseline and an absolute change from Baseline of > 20 points (0-100 scale), OR
  * Improvement in at least two of the following three:
    1. Improvement in pain (KOOS pain subscale) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 points (0-100 scale)
    2. Improvement in function (KOOS function subscale) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 points (0-100 scale)
    3. Improvement in patient's global assessment defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 mm (0-100 scale)
Change from baseline in 4x10 meter fast walk test | Week 9 and week 12
  The 4x10 meter fast walk test (40mFWT) is a physical performance test that quantifies short distance walking performance. The 40mFWT is a measure of walking speed over short distances and changing direction during walking. It is recommended as a performance-based test to assess physical function in people diagnosed with hip or knee OA.
  The participant is asked to walk as quickly but as safely as possible to a mark 10 m away, return, and repeat for a total distance of 40 m. Regular walking aid is allowed and recorded. Time of one trial, with turn time excluded, is recorded and expressed as speed m/s by dividing distance (40 m) by time (s).
Change from baseline in the 30 seconds chair stand test | Week 9 and week 12
  The 30 seconds chair stand test (30sCST) is a physical performance test that quantifies how many sit-to-stand movements an individual is able to perform within 30 seconds. The 30sCST is a measure of balance during functional activities and lower extremity function and strength. It is recommended as a performance-based test to assess physical function in people diagnosed with hip or knee OA.
  From the sitting position in the middle of seat with feet shoulder width apart, flat on the floor, arms crossed at chest, the participant is asked to stand completely up, then sit completely back down, repeatedly for 30 seconds. The total number of complete chair stands (up and down represents one stand) is counted. There is given only one trial. If a full stand is completed at 30 seconds, then this is counted in the total. The same chair is used at all assessments.
Change from baseline in Stair climbing test | Week 9 and week 12
  A stair climbing test (SCT) is a physical performance test that quantifies how fast an individual is able to ascend and descend a flight of stairs in a usual manner. The SCT is a measure of balance during functional activities and lower extremity function and strength. It is recommended as a performance-based test to assess physical function in people diagnosed with hip or knee OA.
  The participant is asked to ascend and descend a flight of stairs in a usual manner, and at a safe and comfortable pace. Use of any walking aid and handrail is permitted and recorded. Total time to ascend and descend steps for one trial is recorded in seconds. The same flight of stairs is used at all assessments.

OTHER OUTCOMES:
Joint fluid aspiration volume | week 9 and 12
  During an ultrasound examination, presence of excess joint fluid will be visualised and, if possible, aspirated by inserting a needle into the joint cavity (under ultrasound guidance). The volume (in ml) of the aspirated fluid will recorded. The ultrasound examination and fluid removal will be conducted by a trained medical doctor (rheumatologist or orthopaedic surgeon).
Change from baseline in swollen knee joint count | week 9 and 12
  An investigator (medical doctor) will examine both knees and record if they are swollen or not based on the presence of palpable effusion. The outcome of the examination will be recorded for each knee as a dichotomous score (present/absent).
Change in current knee pain at treatment visits | Week 1, 2, 3, 4, 5, 6, 7, and 8
  At arrival to each treatment session (education, exercise or injection) we will ask the participants to assess their current knee pain in the target knee a 0-10 points numerical rating scale, with 0 representing "no pain" and 10 representing "worst imaginable pain".
  The assessment is repeated when the participants leave the session and the change on that day is calculated.
Time course pattern of changes from baseline in knee OA symptoms during the treatment period | Weeks 1, 2, 3, 4, 5, 6, 7, and 8
  Assessed by repeated administration of the Knee injury and Osteoarthritis Outcome Score (KOOS)(patient-reported questionnaire) The KOOS consists of 42 items covering five domains, namely, Pain (9 items), Symptoms (7 items), Activities of Daily Living (ADL) (17 items), Sports and Recreation (5 items), and knee-related QoL (4 items). The KOOS adopts a five-point Likert scale scoring system (ranging from 0 (least severe) to 4 (most severe)). A normalized score is calculated for each domain with 0 indicating extreme symptoms and functional impairment and 100 indicating no symptoms and functional impairment.
Time course pattern of changes from baseline in morning knee OA pain | Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9 and 12
  Assessed by repeated administration of a 100 mm analogue scale (VAS) relating to the degree of the patient's perceived averaged morning knee pain during the last week with anchors: 0="No pain" and 100 = "Worst imaginable pain". (patient-reported questionnaire)
Change from baseline in intermittent and constant knee pain | Week 9 and 12
  Assessed by the Measure of Intermittent and Constant Osteoarthritis Pain - ICOAP (patient-reported questionnaire).
Use of acetaminophen and ibuprofen during study participation | Baseline, Week 9 and 12
  Patient reported use of acetaminophen

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, PhD, Study Director — The Parker institute; Henning Bliddal, DMSc, Principal Investigator — The Parker institute
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We will share the IPD, protocol and SAP, but the circumstances and timing has not been decided yet

REFERENCES:
- [Derived] Henriksen M, Christensen R, Kristensen LE, Bliddal H, Bartholdy C, Boesen M, Ellegaard K, Guldberg-Moller J, Hunter DJ, Altman R, Bandak E. Exercise and education vs intra-articular saline for knee osteoarthritis: a 1-year follow-up of a randomized trial. Osteoarthritis Cartilage. 2023 May;31(5):627-635. doi: 10.1016/j.joca.2022.12.011. Epub 2023 Jan 16. PMID 36657659
- [Derived] Henriksen M, Nielsen SM, Christensen R, Kristensen LE, Bliddal H, Bartholdy C, Boesen M, Ellegaard K, Hunter DJ, Altman R, Bandak E. Who are likely to benefit from the Good Life with osteoArthritis in Denmark (GLAD) exercise and education program? An effect modifier analysis of a randomised controlled trial. Osteoarthritis Cartilage. 2023 Jan;31(1):106-114. doi: 10.1016/j.joca.2022.09.001. Epub 2022 Sep 8. PMID 36089229
- [Derived] Bandak E, Christensen R, Overgaard A, Kristensen LE, Ellegaard K, Guldberg-Moller J, Bartholdy C, Hunter DJ, Altman R, Bliddal H, Henriksen M. Exercise and education versus saline injections for knee osteoarthritis: a randomised controlled equivalence trial. Ann Rheum Dis. 2022 Apr;81(4):537-543. doi: 10.1136/annrheumdis-2021-221129. Epub 2021 Nov 29. PMID 34844929
- [Derived] Bandak E, Overgaard AF, Kristensen LE, Ellegaard K, Guldberg-Moller J, Bartholdy C, Hunter DJ, Altman RD, Christensen R, Bliddal H, Henriksen M. Exercise therapy and patient education versus intra-articular saline injections in the treatment of knee osteoarthritis: an evidence-based protocol for an open-label randomised controlled trial (the DISCO trial). Trials. 2021 Jan 6;22(1):18. doi: 10.1186/s13063-020-04952-5. PMID 33407791

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT03843931/SAP_000.pdf